CLINICAL TRIAL: NCT00215124
Title: Phase I - II Safety Study of Filgrastim (Neupogen) to Improve Left Ventricular Function After Severe Acute Myocardial Infarction
Brief Title: A Phase I - II Safety Study of Filgrastim (Neupogen) to Improve Left Ventricular Function After Severe Acute Myocardial Infarction
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5225
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2008-09-19 (Estimated); Status verified 2008-09

CONDITIONS: Acute Myocardial Infarction
MeSH Terms: interventions — Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Filgrastim

SUMMARY:
The objective is to obtain initial information regarding the safety and efficacy of the use of Filgrastim in the setting of acute myocardial infarction.

The secondary objectives are to obtain information regarding the mobilization of relevant stem cell progenitor cells by Filgrastim in this setting and to obtain further clinical information that may be helpful in the assessment of safety and efficacy of this drug as utilized.

It is a one center, randomized, placebo controlled, dose escalation, blinded study. It will be 2:1 randomization with 9 patients total.

Filgrastim 10 mcg/kg/day will be administered SQ for 5 days vs. placebo.

Primary endpoint is death /or myocardial rupture or change in left ventricular ejection fraction from baseline to 30 days.

9 pts. have already completed the first phase of the trial using Filgrastim 5 mcg/kg/day.

ELIGIBILITY:
Inclusion Criteria:

Acute Myocardial Infarction within 6 hours of symptoms

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Death or myocardial rupture at 30 days; change in left ventricular ejection fraction from baseline to 30 days | 30 days

SECONDARY OUTCOMES:
i) Survival through 12 months ii) Re-hospitalization for CHF through 12 months iii) Improvement in LVEF at days 7 and 12 months iv) Infarct wall thickness at 30 days v) Re-infarction within 30 days v | specified above

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Ellis, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Ellis SG, Penn MS, Bolwell B, Garcia M, Chacko M, Wang T, Brezina KJ, McConnell G, Topol EJ. Granulocyte colony stimulating factor in patients with large acute myocardial infarction: results of a pilot dose-escalation randomized trial. Am Heart J. 2006 Dec;152(6):1051.e9-14. doi: 10.1016/j.ahj.2006.09.003. PMID 17161051